CLINICAL TRIAL: NCT04081337
Title: A Randomized, Placebo-Controlled, Parallel-Arm Study to Investigate the Effect of Once-Weekly Tirzepatide on Energy Expenditure and Food Intake in Obese Subjects
Brief Title: A Study to Measure Energy Expenditure and Food Intake in Participants With Obesity Using Tirzepatide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17092; I8F-MC-GPGU (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo once weekly (QW) by Subcutaneous (SC) injection.
  Interventions: Drug: Placebo
- 15 Milligram (mg) Tirzepatide (Experimental): Participants received 15 mg of tirzepatide QW by SC injection.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 15 Milligram (mg) Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This is a study of tirzepatide in participants with obesity. The main purpose is to learn more about how tirzepatide affects the number of calories participants burn and the amount of food they eat. The study lasted for 28 weeks and will include about 21 visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Have body mass index of 30 to 45 kilograms per square meter (kg/m²), inclusive
* Have a stable body weight in the past 1 month prior to screening
* Willing and agreeable to commit to the duration of the study and undergo study procedures as instructed by the clinic staff

Exclusion Criteria:

* Have undergone gastric bypass or bariatric surgery
* Have a diagnosis of type 2 diabetes
* Have a history or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data
* Have received prescription drugs or over the counter drugs that promote weight loss in the past 6 months prior to screening
* Have any lifetime history of a suicide attempt
* Patient Health Questionnaire-9 (PHQ-9) score of 15 or more at screening
* Positive responses to selected items on the Columbia Suicide Severity Rating Scale (C-SSRS)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Measure Food and Calorie Consumption in Very Overweight Participants Using Tirzepatide — https://trials.lillytrialguide.com/en-US/trial/1nfPN3HbtLj7FPbvr6zfwo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 15 Milligram (mg) Tirzepatide
Started | 28 | 27
Received at Least One Dose of Study Drug | 28 | 27
Completed | 24 | 24
Not Completed | 4 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received placebo QW by SC injection.
- 15 mg Tirzepatide: Participants received 15 mg of tirzepatide QW by SC injection.
- Total: Total of all reporting groups
Arm/Group | Placebo | 15 mg Tirzepatide | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (10.7) | 45.5 (9.8) | 46.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 11 | 23
  White | 15 | 14 | 29
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 18 in Sleep Metabolic Rate (SMR)
Description: SMR was measured using whole-room indirect calorimetry (respiratory chamber). Change from Baseline to Week 18 in SMR was evaluated. Least square (LS) mean was determined by analysis of covariance (ANCOVA) model with Baseline, Treatment, Change from Baseline to Week 18 in Fat-Free Mass, Change from baseline to Week 18 in Fat Mass and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and had evaluable data for SMR.
Measure: Least Squares Mean (Standard Error); unit: kilocalories per day (kcal/day)
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 24 | 21
kilocalories per day (kcal/day) | -154.36 (19.69) | -134.68 (21.62)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p = 0.5733, ANCOVA; LS Mean Difference = 19.68, 95% CI 2-sided [-50.36 to 89.72]

2. Secondary Outcome: Change From Baseline to Week 18 in Food Intake During Ad Libitum Meal
Description: Ad libitum lunch and dinner were provided. The sum of the caloric breakdown (carbohydrates, protein, and fats) was calculated from the respective nutritional information of the food items. LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and had evaluable data for food Intake during ad libitum meal.
Measure: Least Squares Mean (Standard Error); unit: kilocalories (kcal)
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 24 | 24
kilocalories (kcal) | -58.57 (82.29) | -914.51 (82.29)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -855.94, 95% CI 2-sided [-1090.87 to -621.02]

3. Secondary Outcome: Change From Baseline to Week 18 in 24-hour Energy Expenditure (EE)
Description: 24 hour energy expenditure was measured in a respiratory chamber. LS mean was determined by ANCOVA model with Baseline, Treatment, Change from Baseline to Week 18 in Fat-Free Mass, Change from baseline to Week 18 in Fat Mass and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and who had evaluable data for 24-hour EE.
Measure: Least Squares Mean (Standard Error); unit: kcal/day
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 24 | 21
kcal/day | -296.85 (27.67) | -300.07 (30.44)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p = 0.9481, ANCOVA; LS Mean Difference = -3.22, 95% CI 2-sided [-102.65 to 96.20]

4. Secondary Outcome: Change From Baseline to Week 18 in 24 Hour Respiratory Quotient (RQ)
Description: Respiratory quotient was calculated as the ratio of carbon dioxide production to oxygen consumption as measured in a metabolic chamber for 24 continuous hours. Ratio of total carbon dioxide production (VCO2)/total oxygen consumption (VO2), from baseline to Week 18 was evaluated. 24-hour RQ = total VCO2 [Liter/24hour] / total VO2 [Liter/24hour]. LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and who had evaluable data for 24-hour RQ.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 24 | 21
Ratio | 0.005 (0.005) | -0.030 (0.006)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.034, 95% CI 2-sided [-0.051 to -0.018]

5. Secondary Outcome: Change From Baseline to Week 18 in Sleep RQ
Description: Sleep RQ is defined as the ratio of VCO2 to VO2 during sleep time points. Change from baseline to Week 18 in sleep RQ is presented. LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and who had evaluable data for sleep RQ.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 24 | 21
ratio | -0.001 (0.006) | -0,028 (0.006)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p = 0.0031, ANCOVA; LS Mean difference = -0.028, 95% CI 2-sided [-0.045 to -0.010]

6. Secondary Outcome: Change From Baseline to Week 18 in Duration of Periods With RQ<0.80
Description: RQ<0.80 is defined as the cut point for high lipid oxidation of RQ; lipid oxidation will be calculated and corrected for protein oxidation; the total number of minutes with RQ <0.80, termed "lipid oxidation duration," during each 23-hour measurement period will be recorded; protein oxidation will be determined from urine nitrogen that will be collected during 2 periods for each calorimeter day. LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and who had evaluable data for duration of periods with RQ<0.80.
Measure: Least Squares Mean (Standard Error); unit: minute
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 24 | 21
minute | 2.55 (43.97) | 254.44 (47.14)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p = 0.0004, ANCOVA; LS Mean difference = 251.89, 95% CI 2-sided [119.09 to 384.69]

7. Secondary Outcome: Change From Baseline to Week 18 in Fat, Protein, and Carbohydrate Oxidation
Description: Change from Baseline to Week 18 in Fat, Protein, and Carbohydrate Oxidation is presented.
  * Protein Oxidation = 6.25*[urinary nitrogen]
  * Fat Oxidation = 1.689*[total oxygen consumption (VO2)] - 1.689*[total carbon dioxide production (VCO2)] - 0.324*[protein oxidation]
  * Carbohydrate Oxidation = 4.113*[VCO2] - 2.907*[VO2] - 0.375*[protein oxidation].
  Adjusted oxidation is calculated using the formula, Adjusted oxidation rate (g/day) = oxidation rate (g/day) / 24-hour Energy Expenditure) x 1000 (kcal/day).
  LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and who had evaluable data for fat, protein, and carbohydrate oxidation.
Measure: Least Squares Mean (Standard Error); unit: gram/day
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 24 | 21
gram/day
  Adjusted protein oxidation | -0.14 (1.23) | -7.00 (1.32)
  Adjusted fat oxidation | -1.64 (2.15) | 12.83 (2.30)
  Adjusted carbohydrate oxidation | 4.23 (4.24) | -22.42 (4.54)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; For Adjusted protein oxidation; Test type: Superiority; p = 0.0005, ANCOVA; LS Mean difference = -6.87, 95% CI 2-sided [-10.51 to -3.22]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; For Adjusted fat oxidation; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean difference = 14.48, 95% CI 2-sided [8.02 to 20.93]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Adjusted carbohydrate oxidation; Test type: Superiority; p = 0.0001, ANCOVA; LS Mean difference = -26.64, 95% CI 2-sided [-39.46 to -13.83]

8. Secondary Outcome: Change From Baseline to Week 18 in Body Weight (BW)
Description: Change from baseline in BW through Week 18 in participants were presented. LS mean was determined by mixed measures repeated model (MMRM) model with Baseline, Treatment, Time, Treatment*Time, Participant and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and who had evaluable data for body weight.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 25 | 24
kilogram (kg) | -8.26 (0.90) | -16.73 (0.92)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean difference = -8.47, 95% CI 2-sided [-11.04 to -5.90]

9. Secondary Outcome: Change From Baseline to Week 18 in Body Fat-Free Mass
Description: Change from baseline to Week 18 in body fat free mass is presented. Body fat free mass was measured using dual energy X-ray absorptiometry (DXA) measurements. LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and who had evaluable data for body fat-free mass.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 24 | 24
kg | -1.64 (0.36) | -5.73 (0.36)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean difference = -4.08, 95% CI 2-sided [-5.12 to -3.05]

10. Secondary Outcome: Change From Baseline to Week 18 in Body Fat Mass
Description: Change from baseline to Week 18 in body fat mass is presented. Body fat mass was measured using DXA measurements. LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and who had evaluable data for body fat mass.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 24 | 24
kg | -6.75 (0.65) | -11.83 (0.65)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean difference = -5.08, 95% CI 2-sided [-6.93 to -3.22]

11. Secondary Outcome: Change From Baseline to Week 18 in Percentage of Body Fat Mass
Description: The total body fat mass was measured in kilograms (kg) using DXA scanning. Change from baseline to week 18 in percentage of body fat mass is reported. LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and who had evaluable data for percentage of body fat mass.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 24 | 24
Percentage | -3.12 (0.36) | -4.26 (0.36)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p = 0.0304, ANCOVA; LS Mean Difference = -1.14, 95% CI 2-sided [-2.16 to -0.11]

12. Secondary Outcome: Change From Baseline to Week 18 in Lipid Metabolism Parameters
Description: Change in Lipid Metabolism Parameters from baseline (week 0) to week 18 is evaluated. Triglyceride, Very low density lipoprotein (VLDL), High density lipoprotein (HDL) cholesterol and free fatty acids values were reported. Results below presents Area under the Curve (AUC) during standardized mixed-meal tolerance test (sMMTT). LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and who had evaluable data for lipid metabolism parameters.
Measure: Least Squares Mean (Standard Error); unit: millimole hour per liter (mmol.h/L)
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 23 | 23
millimole hour per liter (mmol.h/L)
  Triglyceride | -0.69 (0.27) | -2.52 (0.27)
  VLDL cholesterol | -0.32 (0.12) | -1.16 (0.12)
  HDL cholesterol | 0.20 (0.18) | -0.33 (0.18)
  Free fatty acid | -0.09 (0.08) | 0.35 (0.08)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; For Triglyceride; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean difference = -1.83, 95% CI 2-sided [-2.60 to -1.06]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; For VLDL; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean difference = -0.84, 95% CI 2-sided [-1.19 to -0.48]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; For HDL; Test type: Superiority; p = 0.0436, ANCOVA; LS Mean difference = -0.53, 95% CI 2-sided [-1.05 to -0.02]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; For Free fatty acid; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = 0.45, 95% CI 2-sided [0.23 to 0.66]

13. Secondary Outcome: Change From Baseline to Week 18 in Fasting Insulin Resistance
Description: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) is a test that uses a simultaneous fasting blood glucose test and fasting insulin test to accurately estimate the degree of insulin resistance (IR) and β-cell function (the cells of the pancreas that produce insulin).
  HOMA-IR= [Fasting glucose (mmol/L) x (fasting insulin (picomoles per liter {pmol/L})/6)] / 22.5. LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18 during standardized mixed meal tolerance test
Population: All randomized participants who received at least one dose of study drug and who had evaluable HOMA-IR data.
Measure: Least Squares Mean (Standard Error); unit: index
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 23 | 19
index | -0.37 (0.12) | -0.34 (0.14)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p = 0.8762, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.34 to 0.40]

14. Secondary Outcome: Change From Baseline to Week 18 in Postprandial Insulin Sensitivity
Description: Insulin sensitivity was measured from insulin and glucose levels obtained following standard meal challenge using a modification of the Matsuda index. This was calculated based on data obtained from a 75 g oral glucose tolerance test, as follows: 10,000 divided by the square root of {(fasting glucose X fasting insulin) (total area under the glucose response curve (AUC) 0-4hr)) X total insulin AUC(0-4hr )}. A Matsuda index of <2.5 indicates whole body insulin resistance. A lower Matsuda Index indicates the worst disease state. An increase in the Matsuda Index indicates an improvement in insulin sensitivity (best). A positive change from Baseline indicates improvement and a negative change from Baseline indicates a worsening. Stumvoll and oral glucose insulin sensitivity indexes were also used for measuring the insulin Sensitivity. LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and had evaluable data for matsuda index.
Measure: Least Squares Mean (Standard Deviation); unit: index
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 23 | 23
index | 1.43 (0.94) | 4.92 (0.94)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p = 0.0126, ANCOVA; LS Mean difference = 3.49, 95% CI 2-sided [0.79 to 6.19]

15. Secondary Outcome: Change From Baseline to Week 18 in Postmeal Total Glucose AUC During sMMTT
Description: Total AUC from time zero to 4 hours after start of the meal [AUC0-4 hours]) during sMMTT was evaluated. LS mean was determined by ANCOVA model with Baseline, Treatment and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and had evaluable data for postmeal total glucose AUC during sMMTT.
Measure: Least Squares Mean (Standard Error); unit: millimolar.hour per liter (mmol.h/L)
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 23 | 23
millimolar.hour per liter (mmol.h/L) | -1.73 (0.38) | -3.00 (0.38)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p = 0.0222, ANCOVA; LS Mean Difference = -1.26, 95% CI 2-sided [-2.34 to -0.19]

16. Secondary Outcome: Change From Baseline to Week 18 in Hemoglobin A1c (HbA1c)
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. LS mean was determined by ANCOVA model with Baseline, Treatment, Time, Treatment*Time, Participant and Random Error as variables.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and had evaluable data for HbA1c.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Placebo | 15 mg Tirzepatide
Number analyzed (Participants) | 24 | 24
percentage of glycosylated hemoglobin | -0.04 (0.04) | -0.40 (0.04)
Statistical Analysis 1: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean difference = -0.36, 95% CI 2-sided [-0.48 to -0.23]

ADVERSE EVENTS:
Time Frame: Baseline Through End of Safety Follow-up (Up to 22 Weeks)
Description: All randomized participants who received at least one dose of study drug, regardless of whether they completed all protocol requirements. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly. Frequency threshold for reporting other (not including serious) adverse event is greater than or equal to (≥) 5% in any of the treatment groups.
Groups:
- Placebo: Participants received placebo once weekly by SC injection.
- 15 mg Tirzepatide: Participants received 15 mg of tirzepatide once weekly by subcutaneous injection.
Arm/Group | Placebo | 15 mg Tirzepatide
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/27
Other Adverse Events (participants affected / at risk) | 19/28 | 22/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | 15 mg Tirzepatide (N=27)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=28) | 15 mg Tirzepatide (N=27)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (3) | 3 (8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (9) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (5)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 14 (29)
Vomiting (Gastrointestinal disorders) | 3 (4) | 7 (8)
Injection site reaction (General disorders) | 0 (0) | 10 (31)
Pain (General disorders) | 2 (2) | 0 (0)
Corona virus infection (Infections and infestations) | 4 (4) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 9 (10) | 6 (6)
Metrorrhagia (Reproductive system and breast disorders) | 0/24 (0) | 2/22 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT04081337/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT04081337/SAP_001.pdf